CLINICAL TRIAL: NCT07160725
Title: A Phase 1/2a, First-in-human, Open-label Study of BMS-986517 as Monotherapy in Adult Participants With Advanced Solid Tumors
Brief Title: A Phase 1/2a, First-in-human, Study of BMS-986517 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA254-0001; EU CTR (Other: 2025-522203-23); WHO (Other: U1111-1322-1627)
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumours

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 (Experimental)
  Interventions: Drug: BMS-986517
- Part 2: Cohort A (Experimental)
  Interventions: Drug: BMS-986517
- Part 2: Cohort B (Experimental)
  Interventions: Drug: BMS-986517
- Part 2: Cohort C (Experimental)
  Interventions: Drug: BMS-986517

INTERVENTIONS:
Drug: BMS-986517 — Specified dose on specified days

SUMMARY:
A phase 1/2a, open-label, first-in-human study mainly aimed to evaluate the safety and tolerability of BMS-986517 in participants with solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Participants must have an ECOG performance status of 0 to 1.
* Participants must have measurable disease by RECIST v1.1 (radiologically measured by the Investigator).
* Participants must have documented histologically or cytologically confirmed advanced, unresectable/metastatic solid tumors, including NSCLC, HNSCC, TNBC, and HR+/HER2- breast cancer.

Exclusion Criteria:

* Participants must not have untreated CNS metastases. Participants are eligible if CNS metastases have been treated and do not require immediate treatment or have been treated and have neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment).
* Participants must not have concurrent malignancy (present during Screening) requiring treatment or history of prior malignancy active within 2 years prior to treatment assignment.
* Participants must not have history of serious recurrent infections.
* Participants must not have impaired cardiac function or history of severe heart disease.
* Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AE) | Up to approximately 2 years
Number of Participants with Serious Adverse Events (SAE) | Up to approximately 2 years
Number of Participants with AEs meeting protocol-defined Dose-limiting Toxicities (DLTs) criteria | Up to Day 21
  For part 1 only
Number of Participants with AEs Leading to Discontinuation | Up to approximately 2 years
Number of Participants with AEs Leading to Deaths | Up to approximately 2 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Assessed by RECIST v1.1 per investigator assessment | Up to approximately 3 years
Duration of Response (DOR) Assessed by RECIST v1.1 per investigator assessment | Up to approximately 3 years
Maximum Plasma Concentration (Cmax) | Up to approximately 2 years
Time to Reach Maximum Plasma Concentration (Tmax) | Up to approximately 2 years
Area Under Curve (AUC) | Up to approximately 2 years
Total anti-drug antibodies (ADAs) | Up to approximately 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (19):
- United States (9):
  - Local Institution - 0033, Irvine, California
  - Local Institution - 0002, Los Angeles, California
  - Local Institution - 0021, Orange, California
  - Local Institution - 0008, Pittsburgh, Pennsylvania
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - START - Dallas Fort Worth, Fort Worth, Texas
  - START San Antonio, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
  - Local Institution - 0028, Seattle, Washington
- Denmark (3):
  - Herlev and Gentofte Hospital, Copenhagen, Capital Region
  - Odense Universitetshospital, Odense, Region Syddanmark
  - Copenhagen University Hospital Rigshospitalet, Copenhagen
- National Cancer Center Hospital, Chuo-ku, Tokyo, Japan
- Spain (6):
  - Local Institution - 0026, Málaga, Andalusia
  - Local Institution - 0022, Badalona, Barcelona [Barcelona]
  - Local Institution - 0024, Barcelona, Barcelona [Barcelona]
  - Local Institution - 0025, Pamplona, Navarre
  - Local Institution - 0027, Madrid
  - Local Institution - 0023, Madrid

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07160725.html